CLINICAL TRIAL: NCT00129883
Title: Prevention of Antimicrobial Resistance in Hospitals: Promoting Appropriate Use of Antibiotics in Hospital Departments of Internal and Pulmonary Medicine
Brief Title: Adherence to Guidelines for Antibiotic Use in Respiratory Infections at Hospitals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Educational/Counseling/Training
Other Study IDs: AGAR-2001-1; ZonMw grant no. 2300.0024
Record Dates: First submitted 2005-08-11; First posted 2005-08-12 (Estimated); Last update posted 2005-09-27 (Estimated); Status verified 2002-08

CONDITIONS: Pneumonia; Chronic Bronchitis; COPD
Keywords: quality of care; antibiotic use; intervention; lower respiratory tract infections; Community acquired Pneumonia; Acute Exacerbation of Chronic Bronchitis or COPD
MeSH Terms: conditions — Pneumonia; Bronchitis, Chronic; Pulmonary Disease, Chronic Obstructive; Community-Acquired Pneumonia

INTERVENTIONS:
Behavioral: Professional education
Behavioral: Implementation of a Critical Care Pathway
Behavioral: Professional audit and feedback
Behavioral: Process analysis and redesign

SUMMARY:
The purpose of this study is to test a strategy to improve the quality of antibiotic use in lower respiratory tract infections (LRTIs) at hospitals. Therefore, a multifaceted intervention strategy is compared to a control strategy and the effectiveness and feasibility of the intervention is assessed.

DETAILED DESCRIPTION:
Improving processes of care in patients with hospital LRTI has been related to better patient outcome. Inappropriate use of antibiotics has contributed to the emergence and spread of drug-resistant micro organisms and increased treatment costs. International guidelines provide recommendations for the initial evaluation and management of LRTI, including advice on judicious antibiotic therapy. Nonetheless, studies have demonstrated a wide variability in adherence to these guidelines.

To implement key recommendations in clinical practice, various strategies have been used, with mixed results. Perhaps the most important aspect of choosing a potentially effective intervention is that the choice of intervention should be based upon assessment of potential barriers in the target group. Many intervention studies are flawed by failing to control for secular trends.

The investigators performed a cluster randomised controlled trial, to study the effect of a multifaceted intervention strategy on the quality of antibiotic use for LRTI. Their intervention was tailored to the areas most in need for improvement and took perceived barriers in the target group into consideration at the individual hospital level.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to a respiratory care or internal medicine ward with community-acquired pneumonia or acute exacerbation of chronic bronchitis or chronic obstructive pulmonary disease (COPD)

Exclusion Criteria:

* Recent (< 30 days) admission for LRTI
* Patients with underlying immunodeficiency (HIV infection, neutropenia, treatment with immunomodulating drugs, active hematological malignancies, anatomical or functional asplenia and hypogammaglobulinemia)
* Patients already on treatment with antibiotics for another culture proven infection at the time of admission
* Patients from nursing homes
* Patients who had been transferred to another hospital or ICU and patients who had died within 24 hours of admission
* Patients with very poor prognosis (life expectancy < 2 weeks on admission).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000
Dates: Start 2002-09; Study Completion 2005-04

PRIMARY OUTCOMES:
adherence to key quality indicators for antibiotic use in lower respiratory tract infections (indicators were developed from current [inter]national guideline recommendations and a systematic review of the literature)

SECONDARY OUTCOMES:
cost
process evaluation: how well was the intervention performed
length of hospital stay
in-hospital mortality
Intensive Care Unit (ICU)-transfer
30 day re-admission rate

CONTACTS AND LOCATIONS:
Overall Officials: Marlies E Hulscher, MSc, PhD, Principal Investigator — Centre for Quality of Care Research, Radboud University Nijmegen Medical Centre; Richard P Grol, MSc, PhD, Study Director — Centre for Quality of Care Research, Radboud University Nijmegen Medical Centre; Jos WM van der Meer, MD, PhD, Study Director — Department of General Internal Medicine, Radboud University Nijmegen Medical Centre
Locations (7):
- Netherlands (7):
  - Gelre Ziekenhuizen, Apeldoorn
  - Deventer Ziekenhuis, Deventer
  - Ziekenhuis Gelderse Vallei, Ede
  - Bernhoven Ziekenhuis, Oss
  - Bernhoven Ziekenhuis, Veghel
  - Maxima Medisch Centrum, Veldhoven
  - Vie Curi Medisch Centrum, Venlo

REFERENCES:
- See also: website of Centre for Quality of Care Research, department of the Radboud University Nijmegen Medical Centre, where this study was carried out — http://www.wokresearch.nl